CLINICAL TRIAL: NCT00534911
Title: Reducing Depressive Symptoms in Physically Ill Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eva Szigethy, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0606136; NCT00596869 (obsolete NCT alias)
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Inflammatory Bowel Disease; Depression
Keywords: Depression; Physical Illness; Inflammatory Bowel Disease; Cognitive Behavioral Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Primary & Secondary Control Enhancement Training (PASCET)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Supportive Non-Directive Therapy (SNDT) (Active Comparator): Supportive Non-Directive Therapy
  Interventions: Behavioral: Supportive Non-directive Therapy (SNDT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will receive 12 weeks of CBT designed for youth with IBD. During sessions, participants will learn new ways of thinking (e.g., reconstruction of personal physical illness narratives, coping strategies, social skills) and behaving (e.g., positive activities, family communication, sleep hygiene, relaxation) to improve emotional and physical outcomes. Parent sessions will be provided at the beginning, middle, and end of the treatment to improve family understanding and communication about the physical illness and about risks of developing depression. There will also be 6-month booster sessions during follow-up.
  Other Name: Primary and secondary coping enhancement training (PASCET)
  Arms: Cognitive Behavioral Therapy
Behavioral: Supportive Non-directive Therapy (SNDT) — SNDT is a 12-week non-directive therapeutic intervention. Participants will receive social support and quality information about the warning signs and risk factors for depression. Parent sessions will be provided at the beginning, middle, and end of the treatment to improve family understanding and communication about the physical illness and about risks of developing depression. There will also be 6-month booster sessions during follow-up.
  Arms: Supportive Non-Directive Therapy (SNDT)

SUMMARY:
Children and adolescents with inflammatory bowel disease (IBD) have high rates of depressive symptoms and more trouble with daily functioning than those without physical illness. The proposed study will investigate if cognitive behavioral therapy (CBT) is better than supportive therapy (SNDT) in reducing emotional distress and improving functioning in youth ages 9-17 with Crohn's disease or Ulcerative Colitis and depression. This study will also assess the effect of CBT on IBD-related factors such as disease severity, medication adherence, and physical-health related quality of life.

Hypothesis

- Individuals who receive CBT will show more improvement than individuals who receive SNDT.

DETAILED DESCRIPTION:
Children and adolescents with inflammatory bowel disease (IBD) have high rates of depressive symptoms and more trouble with daily functioning than those without physical illness. Furthermore, the medications used to treat IBR, such as steroids, may induce depression. The proposed study will investigate if cognitive behavioral therapy (CBT) is better than supportive therapy (SNDT) in reducing emotional distress and improving functioning in youth ages 9-17 with Crohn's disease and depression. This study will also be the first to assess the effect of CBT on IBD-related factors such as disease severity, medication adherence, and physical-health related quality of life.

Participants will be carefully evaluated for depression and those who have clinically significant depression will be randomly assigned to either CBT designed for youth with IBD or supportive therapy sessions. Youth in the CBT group will learn new ways of thinking and acting to reduce symptoms of depression focused on the reconstruction of negative or hopeless physical illness narratives. Parents in the CBT group will participate in three family sessions designed to improve family understanding and communication about the physical illness and about risks for developing depression. Children in the supportive therapy condition will receive social support and information about IBD and depression similar to what they would likely receive from social workers in their pediatric medical clinic. Because emotional difficulties such as the experience of depressive symptoms have been linked with the severity and course of IBD symptoms, this information may enable parents to better help their child cope with his/her physical illness. In addition, participants in both groups may experience reduced depression and improved quality of life.

It is predicted that those in the CBT group will benefit by learning effective strategies for coping with IBD and depression, enhancing their social skills, and improving family communication skills while those in the supportive therapy group will benefit by receiving social support and useful information. The proposed study will help determine which psychosocial approach is of greater benefit for depressed youth with IBD and provide a model for integrating behavioral treatment to decrease both emotional and IBD-related suffering into the comprehensive medical care for IBD in the pediatric population.

Aim 1(primary) Are there differences between the two types of therapy in terms of improving depression.

Aim 2 (secondary) Are there differences between the two types of therapy in terms of improving IBD activity, quality of life, and medication adherence? Aim 3) (secondary) Are there differences between the two types of therapy in terms of improving sleep and pain? Aim 4) (exploratory) Are anxiety, steroid use, and gender moderators of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

Step 1:

* ages 9 to 17 inclusive
* capable of completing CDI
* meeting diagnostic criteria for CD (the date of diagnosis = date of the first diagnostic test confirming CD)
* absence of mental retardation by history
* having at least one appointment at the GI clinic (this will include patients followed in these clinics as well as those seeking consultation)

Step 2:

* CDI or CDI-P greater than or equal to 10 at Step 1.
* ages between 9-17 inclusive
* having CD

Exclusion Criteria:

* history or current episode of bipolar disorder, eating disorder, or psychotic disorder by DSM-IV criteria
* mental retardation by history
* antidepressant medications within one month of assessment
* suicidality with plan or of severity requiring immediate psychiatric hospitalization or significant act involving intentional self-harm (e.g., cutting or overdose, resulting in medical attention)
* unacceptable risk for dangerousness to others as indicated by homicidal (or other violent) ideation, intent or plan or action, or use of illegal weapons
* current pregnancy by history
* substance abuse by history within one month of enrollment other than nicotine dependence
* current treatment with CBT or failure of previous CBT trial for depression judged adequate by at least 12 treatment sessions over a period of less than 1 year conducted by an appropriately trained mental health provider using a manual
* if currently receiving other psychotherapy modalities willingness to suspend treatment for 12-week acute treatment phase of study

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2007-09; Primary Completion 2013-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CDRS at 3 months | Month 0, Month 3
  Change in Child Depression Rating Scale (CDRS) score from month 0 assessment to three month assessment.

SECONDARY OUTCOMES:
Change from baseline in KSADS diagnosis at 3 months | Month 0, Month 3
  Remission of depressive episode as measured by Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS) from month 0 assessment to 3 month assessment.

OTHER OUTCOMES:
Pediatric Crohns Disease Index | Month 0, Month 3
  Clinician rated instrument of IBD activity which includes symptoms and objective lab results.
Pediatric Ulcerative Colitis Index | Month 0, Month 3
  Clinician rated instrument of gastrointestinal symptoms.
IMPACT 3 | Month 0, Month 3
  Health-related quality life measure. Self report.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD, PhD, Principal Investigator — University of Pittsburgh/ Children's Hospital of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital-Boston, Boston, Massachusetts
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Keerthy D, Youk A, Srinath AI, Malas N, Bujoreanu S, Bousvaros A, Keljo D, DeMaso DR, Szigethy EM. Effect of Psychotherapy on Health Care Utilization in Children With Inflammatory Bowel Disease and Depression. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):658-664. doi: 10.1097/MPG.0000000000001207. PMID 27035372
- [Derived] Szigethy E, Youk AO, Gonzalez-Heydrich J, Bujoreanu SI, Weisz J, Fairclough D, Ducharme P, Jones N, Lotrich F, Keljo D, Srinath A, Bousvaros A, Kupfer D, DeMaso DR. Effect of 2 psychotherapies on depression and disease activity in pediatric Crohn's disease. Inflamm Bowel Dis. 2015 Jun;21(6):1321-8. doi: 10.1097/MIB.0000000000000358. PMID 25822010
- [Derived] Srinath A, Young E, Szigethy E. Pain management in patients with inflammatory bowel disease: translational approaches from bench to bedside. Inflamm Bowel Dis. 2014 Dec;20(12):2433-49. doi: 10.1097/MIB.0000000000000170. PMID 25208108
- [Derived] Szigethy E, Bujoreanu SI, Youk AO, Weisz J, Benhayon D, Fairclough D, Ducharme P, Gonzalez-Heydrich J, Keljo D, Srinath A, Bousvaros A, Kirshner M, Newara M, Kupfer D, DeMaso DR. Randomized efficacy trial of two psychotherapies for depression in youth with inflammatory bowel disease. J Am Acad Child Adolesc Psychiatry. 2014 Jul;53(7):726-35. doi: 10.1016/j.jaac.2014.04.014. Epub 2014 May 10. PMID 24954822